CLINICAL TRIAL: NCT04670211
Title: Observational Comparison of Tooth-borne, Bone-borne and Hybrid Distraction Following SARPE.
Acronym: SARPE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: ZOL (Other)
Responsible Party: Principal Investigator, Oliver da Costa Senior, dr. Oliver da Costa Senior (principle investigator), ZOL
Other Study IDs: CTU2020095
Record Dates: First submitted 2020-12-01; First posted 2020-12-17 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Malocclusion
Keywords: SARPE; distraction osteogenesis; transverse maxillary hypoplasia
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Tooth-borne distractor: Maxillary distraction with the use of a tooth-borne distractor following Surgically-assisted Rapid Palatal Expansion (SARPE) surgery.
  Interventions: Device: maxillary distractor
- Bone-borne distractor: Maxillary distraction with the use of a bone-borne distractor following Surgically-assisted Rapid Palatal Expansion (SARPE) surgery.
  Interventions: Device: maxillary distractor
- Hybrid distractor: Maxillary distraction with the use of a hybrid distractor following Surgically-assisted Rapid Palatal Expansion (SARPE) surgery.
  Interventions: Device: maxillary distractor

INTERVENTIONS:
Device: maxillary distractor — the type of maxillary distractor: tooth-borne, bone-borne or hybrid distractor

SUMMARY:
The investigators will perform a prospective, non-randomized observational study. The aim of this study is to evaluate stability of tooth-borne, bone-borne and hybrid expansion following SARPE by using data collected according to the existing SARPE follow-up protocol. The insights of this study might elucidate the preferred expansion technique and improve surgical technique.

DETAILED DESCRIPTION:
Maxillary transverse discrepancy (MTD) is a difficult deformity to correct. In skeletal immature patients, an orthopedic-orthodontic expansion is the preferred treatment strategy. In case of a skeletal mature patient, a surgical treatment should be considered. A Surgically assisted Rapid Palatal Expansion (SARPE) procedure is a common surgical treatment for MTD in skeletal mature patients. In this procedure the skeletally mature, maxillary sutures are surgically reopened. One week postoperatively, the patient will activate the expander appliance. There are three widely-used expander appliances: tooth-borne, bone-borne and hybrid expanders. The use of the expander appliance is based on surgeon and referring orthodontist's common practice and preference. A tooth-borne expander is an appliance which is supported by the teeth and bridges the palate. A bone-borne expander is surgically placed at the level of the palate during SARPE surgery. Hybrid expansion is a combination of tooth-borne and bone-borne expansion. These appliances progressively widen the maxilla by daily activation of the distractor. The activation is stopped when the surgeon and/or referring orthodontist judge that the maxilla is sufficiently expanded. However, historical research with the use of cast model's and 2D posteroanterior cephalograms suggest that this expansion is not stable. With the emergence of 3D Cone-Beam Computed Tomography (CBCT) and its appliance as standard of care for pre-operative diagnosis and postoperative follow-up, stability and complications can be assessed more accurately. The goal of this study is to prospectively evaluate stability following SARPE, by analyzing the clinical and radiological data collected according to the existing clinical SARPE follow-up protocol. The secondary outcome is to evaluate complications following the three distractors.

ELIGIBILITY:
Inclusion Criteria:

* Maxillary transverse discrepancy
* Skeletal mature patients
* SARPE treatment is indicated

Exclusion Criteria:

* Patients with a syndrome with an influence on head-and-neck morphology (such as Apert, Crouzon syndrome)
* Cleft patients

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing SARPE surgery due to maxillary transverse discrepancy
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Stability | 1 year postoperatively
  Stability of the maxillary expansion following SARPE. The stability will be evaluated by comparing the CBCT imaging which is taken at the time of maximal transversal maxillary expansion with the CBCT taken one year postoperatively. Width between the mesiobuccal cusps of the first molars and width between the cusps of the canines is measured. Moreover the width of the apertura piriformis and between the palatal foramen is examined in order to evaluate skeletal stability. This allows calculation of the dental and skeletal stability following SARPE.

SECONDARY OUTCOMES:
Complications | 1 year postoperatively
  Complications following SARPE surgery are examined. Anamnestic, clinical and radiographic information is examined in order to determine postoperative complications. The following complications can be examined: postoperative bleeding, mucosal infection, maxillary sinus infection, palatal necrosis, oro-antral communication, gingival recession, tooth discoloration, bone resorption, malunion, nonunion, root resorption, loss of teeth, mechanical failure of the distractor, asymmetric expansion, lacrimation.

IPD SHARING:
Plan to Share IPD: Undecided
On request